CLINICAL TRIAL: NCT04684277
Title: Effectiveness of Internet-Based Interventions for Treatment Compliance and Outcomes of Major Depressive Disorder
Brief Title: Internet-Based Interventions for MDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Si Tianmei, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SF2020-2-4113
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Depression; Medication Adherence
MeSH Terms: conditions — Depression; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- antidepressant treatment (Experimental): recieve antidepressant treatment
  Interventions: Drug: antidepressant treatment
- antidepressant treatment combined with Internet-based interventions (Experimental): recieve antidepressant treatment combined with Internet-based interventions
  Interventions: Other: antidepressant treatment combined with Internet-based interventions

INTERVENTIONS:
Drug: antidepressant treatment — depression recieve antidepressant treatment
  Arms: antidepressant treatment
Other: antidepressant treatment combined with Internet-based interventions — depression recieve antidepressant treatment combined with Internet-based interventions
  Arms: antidepressant treatment combined with Internet-based interventions

SUMMARY:
The acute and remission depression patients of 18-65 years old were recruited. At the time of enrollment, the demographic, symptomatic, neuropsychological and medication adherence data was collected. After the completion of the baseline assessment and examination, the patients were given antidepressant treatment or antidepressant treatment combined with Internet-based interventions. Clinical evaluation was performed at 1, 3 months (acute patients) and 6, 12 months (remission patients) after treatment, including the medication adherence, therapeutic efficacy, recurrence rate and functional rehabilitation. Through above work, this research is expected to provide clinicians with a set of Internet generalized technologies to improve the compliance and clinical outcomes of patients with depression, and to provide patients with treatment and management of the entire disease cycle.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years old, acute (HAMD17 > 17) and remission (HAMD17 < 8) depression

Exclusion Criteria:

* other mental illnesses, serious somatic illnesses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
HAMD17 reduction ratio | 3 months
  The difference of HAMD17 reduction ratio between the two groups was compared
recurrence rate | 12 months
  The difference of recurrence rate between the two groups was compared

CONTACTS AND LOCATIONS:
Overall Officials: Tianmei Si, PhD, Principal Investigator — Institute of mental health, Peking University
Locations (1):
- Yunai Su, Beijing, China

IPD SHARING:
Plan to Share IPD: No